CLINICAL TRIAL: NCT00006465
Title: Phase I Study of Oxaliplatin (NSC# 266046), Irinotecan, and Capecitabine in Patients With Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU5Y99; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-5Y99 (Other: Case Comprehensive Cancer Center); NCI-370
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine — Patients receive oral capecitabine twice daily on days 1-5 weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan and capecitabine until the maximum tolerated dose(MTD).
Drug: irinotecan hydrochloride — Patients receive irinotecan IV over 30 minutes once weekly for 4 weeks (one hour after oxaliplatin). Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan and capecitabine until the maximum tolerated dose(MTD).
  Other Names: camptothecin-11; irinotecan; irinotecan HCl
Drug: oxaliplatin — Patients receive oxaliplatin IV over 2 hours. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Other Names: diaminocyclohexane oxalatoplatinum; oxalatoplatin; oxalatoplatinum

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of irinotecan and capecitabine when given in combination with a fixed dose of oxaliplatin in patients with advanced solid tumors.
* Determine the pharmacokinetic parameters of this regimen in these patients.
* Determine the antitumor response of these patients treated with this regimen.

OUTLINE: This is a dose-escalation study of irinotecan and capecitabine.

Patients receive oxaliplatin IV over 2 hours followed 1 hour later by irinotecan IV over 30 minutes once weekly for 4 weeks. Patients also receive oral capecitabine twice daily on days 1-5 weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 9-15 patients will be accrued for this study within 9-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor not amenable to curative surgery, radiotherapy, or chemotherapy
* Bidimensionally measurable or evaluable disease
* No brain metastases or primary brain tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 4,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT less than 2 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* No known hypersensitivity to fluorouracil

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin and carmustine) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior large-field radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-12; Primary Completion 2003-11 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and dose-limiting toxicity of irinotecan and capecitabine when given in combination with a fixed dose of oxaliplatin in patients with advanced solid tumors. | Treatment cycle is four weeks, repeated every six weeks in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Krishnamurthi SS, Brell JM, Hoppel CL, Egorin MJ, Weaver KC, Li X, Ingalls ST, Zuhowski EG, Schluchter MD, Dowlati A, Cooney MM, Gibbons J, Overmoyer BA, Ivy SP, Remick SC. Phase I clinical and pharmacokinetic study of oxaliplatin, irinotecan and capecitabine. Cancer Chemother Pharmacol. 2009 Feb;63(3):441-50. doi: 10.1007/s00280-008-0754-2. Epub 2008 Apr 15. PMID 18414865